CLINICAL TRIAL: NCT03926533
Title: Telehealth-Enhanced Patient-Oriented Recovery Trajectory After Intensive Care Pilot Feasibility Study
Brief Title: TelePORT Pilot Study
Acronym: TelePORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: American Association of Critical Care Nurses (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Leanne M Boehm, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 190790
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Critical Illness; Acute Respiratory Distress Syndrome; Septic Shock
Keywords: Post-Intensive Care Syndrome
MeSH Terms: conditions — Critical Illness; Respiratory Distress Syndrome; Shock, Septic; postintensive care syndrome | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth ICU Recovery Program (Experimental): Components of the ICU RC telehealth visit will be structured parallel to what is done during a typical in-person clinic visit. The telehealth intervention consists of 5 chronological components conducted during two 1.5 hour telehealth clinic visits (the same time required for an in-person visit). Upon completion of the pre-intervention baseline assessment, the study coordinator will contact patients randomized to the intervention arm to schedule the first telehealth visit. Study visits will occur at 3 weeks and 3 months following hospital discharge.
  Interventions: Other: Telehealth
- Standard Recovery Conditions (No Intervention): participants assigned to the standard of care control group will be contacted by the study coordinator to ensure the patient has a primary care and/or specialist appointment scheduled. At this time, patients will also receive an electronic PICS guide for ICU survivors created by the Society of Critical Care Medicine. Patients will be directed to use the information provided in the PICS guide for ICU survivors to connect with resources.

INTERVENTIONS:
Other: Telehealth — Telehealth visits will be conducted from a private telehealth lab room in the Vanderbilt ICU Recovery Center using a live and interactive approach where providers and patients interact and communicate in real-time using Zoom, a secure video-conferencing platform recommended by Vanderbilt Telehealth.
  Arms: Telehealth ICU Recovery Program

SUMMARY:
Although more than 50% of survivors of critical illness experience one or more post-intensive care syndrome (PICS) problems, there are still no validated interventions for the management of PICS. The long-term goal of this study is to develop and refine in-person and telehealth strategies for the delivery of Intensive Care Unit (ICU) recovery care for the treatment of PICS.

DETAILED DESCRIPTION:
The overall objectives in this application are to (a) examine the feasibility of providing telehealth ICU recovery care and (b) determine if ICU recovery care is effective. The central hypothesis is that ICU recovery care improves cognitive, mental health, and physical function of ICU survivors by application of a patient-centered survivorship care plan with targeted interventions to address patient-specific cognitive, mental health, and physical dysfunctions. The rationale for this project is that a determination of the feasibility of telehealth and effectiveness of ICU recovery care in general is likely to offer a strong scientific framework informing the development of new implementation strategies. We will test the central hypotheses by pursuing two specific aims: 1) Test that telehealth ICU recovery care is feasible, and 2) Test the hypothesis that telehealth ICU recovery care compared to standard of care conditions will be more effective for improvement in cognitive, mental health, physical, and global function at 6 months following hospital discharge. To address these aims, we will enroll patients treated for septic shock and acute respiratory distress syndrome in the medical and surgical ICUs at Vanderbilt University Medical Center. Study patients will be randomized 1:1 to either the telehealth ICU recovery care or standard of care groups. We will conduct telehealth ICU recovery care from the Vanderbilt ICU Recovery Center. This ICU survivor clinic relies on the expertise of clinicians from critical care medicine, nursing, pharmacy, neuropsychology, rehabilitation, and case management to assess and manage PICS. Telehealth feasibility measures include appropriateness, acceptability, and implementability. Following telehealth clinic participation at 3 weeks and 3 months after hospital discharge, we will assess participants for cognitive, mental health, physical, and global quality of life outcomes using trained, blinded research personnel at 6 months following hospital discharge. We incorporated PROMIS patient-centered outcome measures into each patient outcome category. This research is significant because it is expected to provide scientific justification for the continued development and implementation of ICU recovery care programs. Ultimately, such knowledge has the potential to improve the quality of life for millions of ICU survivors and their family members.

ELIGIBILITY:
Inclusion Criteria:

* index ICU stay with a diagnosis of sepsis or acute respiratory distress syndrome projected to be discharged alive as these patients are at the highest risk for developing PICS

Exclusion Criteria:

1. no access to computer, electronic device (e.g., tablet, smartphone), and/or internet connection for virtual clinic visit,
2. primary care received outside of VUMC network,
3. hospice care at discharge,
4. substance abuse or psychiatric disorder that prevents independent living,
5. blind, deaf, unable to speak English, or
6. severe dementia prior to index hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Acceptability | 6 months
  participants will complete the 4-item Likert response Acceptability of Intervention Measure (AIM) of perceived intervention acceptability. Items are measured on a 5-point Likert scale (Completely Disagree = 1 Completely Agree = 5 ). Higher scores indicate greater acceptability. Scores are based on calculated mean.
participants will complete the 4-item Likert response Feasibility of Intervention Measure (FIM) | 6 months
  participants will complete the 4-item Likert response Feasibility of Intervention Measure (FIM) of perceived intervention feasibility. Items are measured on a 5-point Likert scale (Completely Disagree = 1 Completely Agree = 5 ). Higher scores indicate greater feasibility. Scores are based on calculated mean.
Appropriateness | 6 months
  participants will complete the 4-item Likert response Intervention Appropriateness Measure (IAM) of perceived intervention appropriateness. Items are measured on a 5-point Likert scale (Completely Disagree = 1 Completely Agree = 5 ). Higher scores indicate greater appropriateness. Scores are based on calculated mean.

SECONDARY OUTCOMES:
cognitive impairment | 6 months
  The MOCA-Blind is a 13-item widely used measure in research to evaluate for cognitive impairment. The MOCA-Blind assesses memory, attention, language, recall, orientation, and abstraction where total test score ranges from 0 (worst) to 22 (best) and a score below 18 is considered abnormal. The PROMIS Cognitive Function Short-Form v2.0 is an 8-item patient-reported outcome measure that assesses patient-perceived changes in mental acuity, verbal and nonverbal memory, concentration, and verbal fluency. Raw scores are converted to a T-score which rescales the raw score into a standardized score with a mean of 50 (+/-10). Higher T-scores indicates higher function.
depression | 6 months
  Depression will be measured using the PROMIS Depression v1.0, an 8-item self-report of negative mood, views of self, social cognition, and decreased positive affect and engagement. Subjects rate each item from 1 (never) to 5 (always) to indicate the degree to which they have experienced the symptom in the past 7 days. Raw scores for PROMIS Depression are converted to a T-score which rescales the raw score into a standardized score with a mean of 50 (+/-10). Higher T-scores indicate greater depression.
physical impairments | 6 months
  PROMIS Physical Function v2.0, a 20-item self-report of physical capability rather than actual performance of physical activities (e.g., dexterity, mobility). Subjects rate each item from 1 (unable to do) to 5 (without any difficulty) for their current capability. Raw scores are converted to a T-score which rescales the raw score into a standardized score with a mean of 50 (+/-10). Higher T-scores indicate better function. Respiratory function will be measured using the St. George Respiratory Questionnaire (SGRQ), a 40-item self-report questionnaire evaluating pulmonary function, symptoms, and the impact on daily life. Scores range from 0 (no impairment) to 80 (maximum health impairment).
QOL | 6 months
  PROMIS Global Short Form v1.1, a 10-item self-reported measure of health-related quality of life. Subjects rate each item from 1 (poor) to 5 (excellent) for their current health and quality of life with the exception of question #10 which rates pain from 0 (no pain) to 10 (worst imaginable pain). Raw scores are converted to a T-score which rescales the raw score into a standardized score with a mean of 50 (+/-10). Higher T-scores indicate better health-related quality of life.
anxiety | 6 months
  Anxiety will be measured using the PROMIS Anxiety v1.0, an 8-item self-report of fear, anxious misery, hyperarousal, and somatic symptoms. Similar to depression, subjects rate each item from 1 (never) to 5 (always) to indicate the degree to which they have experienced the symptom in the past 7 days. Raw scores for PROMIS Anxiety are converted to a T-score which rescales the raw score into a standardized score with a mean of 50 (+/-10). Higher T-scores indicate greater anxiety.
PTSD symptoms will be measured using the PTSD Checklist for DSM-5 (PCL-5) | 6 months
  PTSD symptoms will be measured using the PTSD Checklist for DSM-5 (PCL-5), a 20-item brief screening tool assessing symptoms of PTSD associated with pre-specified traumatic event (i.e., critical illness), corresponds to the DSM-5 diagnostic criteria for PTSD, and has excellent reliability and sensitivity. Subjects rate each item from 1 (not at all) to 5 (extremely) to indicate the degree to which they have been bothered by a particular symptom over the past month. The total possible score ranges from 0-80 with higher scores indicating more severe symptoms and a cut-off of 50 optimal for indicating a probable diagnosis of PTSD.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boehm LM, Danesh V, LaNoue M, Trochez RJ, Jones AC, Kimpel CC, Sevin CM. Factors Influencing Engagement with in-Person Intensive Care Unit Recovery Clinic Services. J Intensive Care Med. 2023 Apr;38(4):375-381. doi: 10.1177/08850666221127154. Epub 2022 Sep 21. PMID 36128790
- [Result] Boehm LM, Danesh V, Eaton TL, McPeake J, Pena MA, Bonnet KR, Stollings JL, Jones AC, Schlundt DG, Sevin CM. Multidisciplinary ICU Recovery Clinic Visits: A Qualitative Analysis of Patient-Provider Dialogues. Chest. 2023 Apr;163(4):843-854. doi: 10.1016/j.chest.2022.10.001. Epub 2022 Oct 13. PMID 36243061
- [Result] Kovaleva MA, Jones AC, Kimpel CC, Lauderdale J, Sevin CM, Stollings JL, Jackson JC, Boehm LM. Patient and caregiver experiences with a telemedicine intensive care unit recovery clinic. Heart Lung. 2023 Mar-Apr;58:47-53. doi: 10.1016/j.hrtlng.2022.11.002. Epub 2022 Nov 15. PMID 36399862
- [Result] Kovaleva MA, Jones AC, Kimpel CC, Lauderdale JL, Sevin CM, Boehm LM. Patients' and Caregivers' Perceptions of Intensive Care Unit Hospitalization and Recovery. Am J Crit Care. 2022 Jul 1;31(4):319-323. doi: 10.4037/ajcc2022945. PMID 35773198
- [Derived] Eaton TL, Danesh V, Jones AC, Kimpel CC, Sevin CM, Su H, Toth KM, Valley TS, Iwashyna TJ, Boehm LM, McPeake J. Clinician and Patient Responses to US Health Insurers' Policies: A Qualitative Study of Higher Risk Patients. Health Serv Res. 2025 Jun;60(3):e14615. doi: 10.1111/1475-6773.14615. Epub 2025 Apr 24. PMID 40275640
- [Derived] Hussain AA, Jones AC, Hosey MM, Kiehl A, Danesh V, McPeake J, Toth K, Eaton TL, Su H, Jackson JC, Boehm LM. Patient-psychologist telemedicine interactions in an intensive care unit recovery clinic: Qualitative secondary analysis. Intensive Crit Care Nurs. 2025 Apr;87:103886. doi: 10.1016/j.iccn.2024.103886. Epub 2024 Nov 21. PMID 39577128
- [Derived] Carter SJ, Lauderdale J, Stollings JL, Sevin CM, Cunningham-Erves J, Kokoy S, Clouse K, Boehm LM. Factors Influencing Influenza and COVID-19 Vaccine Decision-Making in the Post-ICU Period: A Secondary Analysis. CHEST Crit Care. 2023 Dec;1(3):100027. doi: 10.1016/j.chstcc.2023.100027. Epub 2023 Oct 23. PMID 38188262
- [Derived] Danesh V, McDonald AD, McPeake J, Eaton TL, Potter K, Su H, Jackson JC, Boehm LM. Driving decisions after critical illness: Qualitative analysis of patient-provider reviews during ICU recovery clinic assessments. Int J Nurs Stud. 2023 Oct;146:104560. doi: 10.1016/j.ijnurstu.2023.104560. Epub 2023 Jul 4. PMID 37531701
- See also: The ICU Recovery Center at Vanderbilt — https://www.icudelirium.org/the-icu-recovery-center-at-vanderbilt